CLINICAL TRIAL: NCT01908426
Title: A Phase 3, Randomized, Double-blind, Controlled Study of Cabozantinib (XL184) vs Placebo in Subjects With Hepatocellular Carcinoma Who Have Received Prior Sorafenib
Brief Title: Study of Cabozantinib (XL184) vs Placebo in Subjects With Hepatocellular Carcinoma Who Have Received Prior Sorafenib
Acronym: CELESTIAL
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Exelixis (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XL184-309
Record Dates: First submitted 2013-07-23; First posted 2013-07-25 (Estimated); Results first posted 2019-03-01 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Hepatocellular Carcinoma
Keywords: cabozantinib; XL184; liver cancer; hepatocellular carcinoma; tyrosine kinase inhibitor; MET kinase; vascular endothelial growth factor receptor 2 (VEGFR2)
MeSH Terms: conditions — Carcinoma, Hepatocellular; Liver Neoplasms | interventions — cabozantinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cabozantinib (XL184) (Experimental): Cabozantinib (XL184) 60 mg tablet once daily
  Interventions: Drug: Cabozantinib tablets
- Placebo (Placebo Comparator): Oral cabozantinib-matched placebo tablet once daily
  Interventions: Drug: Placebo tablets

INTERVENTIONS:
Drug: Cabozantinib tablets
  Other Names: XL184
  Arms: Cabozantinib (XL184)
Drug: Placebo tablets
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of Cabozantinib (XL184) compared with placebo on overall survival in subjects with advanced hepatocellular carcinoma who have received prior sorafenib.

ELIGIBILITY:
Select Inclusion Criteria:

1. Histological or cytological diagnosis of HCC.
2. The subject has disease that is not amenable to a curative treatment approach.
3. Received prior sorafenib.
4. Progression following at least 1 prior systemic treatment for HCC.
5. Recovery to from toxicities related to any prior treatments.
6. ECOG performance status of 0 or 1.
7. Adequate hematologic and renal function, based upon meeting protocol defined laboratory criteria within 7 days before randomization.
8. Child-Pugh Score of A.
9. Antiviral therapy per local standard of care if active hepatitis B (HBV) infection.
10. Sexually active fertile subjects(male and female)must agree to use medically accepted methods of contraception during the course of the study and for 4 months after the last dose of study treatment.
11. Female subjects of childbearing potential must not be pregnant at screening.

Select Exclusion Criteria:

1. Fibrolamellar carcinoma or mixed hepatocellular cholangiocarcinoma.
2. Receipt of more than 2 prior systemic therapies for advanced HCC.
3. Any type of anticancer agent (including investigational) within 2 weeks before randomization.
4. Radiation therapy within 4 weeks (2 weeks for radiation for bone metastases) or radionuclide treatment within 6 weeks of randomization.
5. Prior cabozantinib treatment.
6. Known brain metastases or cranial epidural disease unless adequately treated with radiotherapy and/or surgery and stable for at least 3 months before randomization.
7. Concomitant anticoagulation, at therapeutic doses, with anticoagulants.
8. Serious illness other than cancer that would preclude safe participation in the study.
9. Subjects with untreated or incompletely treated varices with bleeding or high risk for bleeding.
10. Moderate or severe ascites.
11. Pregnant or lactating females.
12. Diagnosis of another malignancy within 2 years before randomization, except for superficial skin cancers, or localized, low-grade tumors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 707 (Actual)
Dates: Start 2013-09-26; Primary Completion 2017-10-16 (Actual); Study Completion 2021-01-12 (Actual)

CONTACTS AND LOCATIONS:
Locations (91):
- United States (20):
  - Corona, California
  - Los Angeles, California
  - San Diego, California
  - San Francisco, California
  - Gainesville, Florida
  - Atlanta, Georgia
  - Honolulu, Hawaii
  - Chicago, Illinois
  - Burlington, Massachusetts
  - Rochester, Minnesota
  - Kansas City, Missouri
  - St Louis, Missouri
  - Las Vegas, Nevada
  - East Orange, New Jersey
  - New York, New York
  - Valhalla, New York
  - Dallas, Texas
  - San Antonio, Texas
  - Seattle, Washington
  - Spokane, Washington
- Australia (8):
  - Camperdown, New South Wales
  - Concord, New South Wales
  - Darlinghurst, New South Wales
  - Kogarah, New South Wales
  - Westmead, New South Wales
  - Kurralta Park, South Australia
  - Melbourne, Victoria
  - Perth, Western Australia
- Belgium (4):
  - Edegem, Antwerpen
  - La Louvière, Hainaut
  - Ghent, Oost-Vlaanderen
  - Liège
- Canada (3):
  - Calgary, Alberta
  - Toronto, Ontario
  - Saskatoon, Saskatchewan
- France (8):
  - Nice, Alpes-Maritimes
  - Amiens, Somme
  - Créteil, Val-de-Marne
  - Besançon
  - Bordeaux
  - Clermont-Ferrand
  - Lille
  - Lyon
- Germany (7):
  - Esslingen am Neckar, Baden-Wurttemberg
  - Tübingen, Baden-Wurttemberg
  - München, Bavaria
  - Frankfurt am Main, Hesse
  - Magdeburg, Saxony-Anhalt
  - Berlin
  - Freiburg im Breisgau
- Hong Kong, Hong Kong
- Dublin, Ireland
- Italy (10):
  - Bologna, Emilia-Romagna
  - Faenza, Emilia-Romagna
  - Meldola, Emilia-Romagna
  - Rimini, Emilia-Romagna
  - Rome, Lazio
  - Genoa, Liguria
  - Milan, Lombardy
  - Rozzano, Lombardy
  - Palermo, Sicily
  - Padua, Veneto
- Netherlands (3):
  - Maastricht, Limburg
  - Amsterdam, North Holland
  - Leiden, South Holland
- Auckland, North Island, New Zealand
- Poland (3):
  - Olsztyn, Warmian-Masurian Voivodeship
  - Mysłowice
  - Poznan
- Romania (2):
  - Cluj-Napoca, Cluj
  - Brasov
- Singapore, Singapore
- South Korea (5):
  - Goyang, Gyeonggido
  - Busan
  - Seongnam
  - Seoul
  - Suwon
- Spain (5):
  - Elche, Alicante
  - Majadahonda, Madrid
  - Torrejón de Ardoz, Madrid
  - Madrid
  - Zaragoza
- Taiwan (3):
  - Liuying Township, Tainan
  - Taichung
  - Taipei
- Turkey (Türkiye) (2):
  - Edirne
  - Gaziantep
- United Kingdom (4):
  - Metropolitan Borough of Wirral, England
  - Birmingham
  - London
  - Manchester

REFERENCES:
- [Derived] Freemantle N, Mollon P, Meyer T, Cheng AL, El-Khoueiry AB, Kelley RK, Baron AD, Benzaghou F, Mangeshkar M, Abou-Alfa GK. Quality of life assessment of cabozantinib in patients with advanced hepatocellular carcinoma in the CELESTIAL trial. Eur J Cancer. 2022 Jun;168:91-98. doi: 10.1016/j.ejca.2022.03.021. Epub 2022 Apr 26. PMID 35487183
- [Derived] El-Khoueiry AB, Meyer T, Cheng AL, Rimassa L, Sen S, Milwee S, Kelley RK, Abou-Alfa GK. Safety and efficacy of cabozantinib for patients with advanced hepatocellular carcinoma who advanced to Child-Pugh B liver function at study week 8: a retrospective analysis of the CELESTIAL randomised controlled trial. BMC Cancer. 2022 Apr 9;22(1):377. doi: 10.1186/s12885-022-09453-z. PMID 35397508
- [Derived] Kelley RK, Miksad R, Cicin I, Chen Y, Klumpen HJ, Kim S, Lin ZZ, Youkstetter J, Hazra S, Sen S, Cheng AL, El-Khoueiry AB, Meyer T, Abou-Alfa GK. Efficacy and safety of cabozantinib for patients with advanced hepatocellular carcinoma based on albumin-bilirubin grade. Br J Cancer. 2022 Mar;126(4):569-575. doi: 10.1038/s41416-021-01532-5. Epub 2021 Oct 7. PMID 34621044
- [Derived] Trojan J, Mollon P, Daniele B, Marteau F, Martin L, Li Y, Xu Q, Piscaglia F, Zaucha R, Sarker D, Lim HY, Venerito M. Comparative Efficacy of Cabozantinib and Ramucirumab After Sorafenib for Patients with Hepatocellular Carcinoma and Alpha-fetoprotein >/= 400 ng/mL: A Matching-Adjusted Indirect Comparison. Adv Ther. 2021 May;38(5):2472-2490. doi: 10.1007/s12325-021-01700-2. Epub 2021 Apr 6. PMID 33822328
- [Derived] Kelley RK, Ryoo BY, Merle P, Park JW, Bolondi L, Chan SL, Lim HY, Baron AD, Parnis F, Knox J, Cattan S, Yau T, Lougheed JC, Milwee S, El-Khoueiry AB, Cheng AL, Meyer T, Abou-Alfa GK. Second-line cabozantinib after sorafenib treatment for advanced hepatocellular carcinoma: a subgroup analysis of the phase 3 CELESTIAL trial. ESMO Open. 2020 Aug;5(4):e000714. doi: 10.1136/esmoopen-2020-000714. PMID 32847838
- [Derived] Abou-Alfa GK, Meyer T, Cheng AL, El-Khoueiry AB, Rimassa L, Ryoo BY, Cicin I, Merle P, Chen Y, Park JW, Blanc JF, Bolondi L, Klumpen HJ, Chan SL, Zagonel V, Pressiani T, Ryu MH, Venook AP, Hessel C, Borgman-Hagey AE, Schwab G, Kelley RK. Cabozantinib in Patients with Advanced and Progressing Hepatocellular Carcinoma. N Engl J Med. 2018 Jul 5;379(1):54-63. doi: 10.1056/NEJMoa1717002. PMID 29972759

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First patient enrolled: 26 September 2013, Data cut-off date: 01 June 2017
Groups:
- Cabozantinib (XL184): Cabozantinib (XL184) 60 mg tablet once daily
  Cabozantinib tablets
- Placebo: Oral cabozantinib-matched placebo tablet once daily
  Placebo tablets
Period: Overall Study
Arm/Group | Cabozantinib (XL184) | Placebo
Started | 470 | 237
Completed | 73 | 26
Not Completed | 397 | 211
Not completed — Adverse Event | 98 | 11
Not completed — Clinical Deterioration | 72 | 38
Not completed — Lack of Efficacy | 3 | 0
Not completed — Lost to Follow-up | 0 | 1
Not completed — Physician Decision | 3 | 3
Not completed — Withdrawal by Subject | 11 | 6
Not completed — Progressive Disease | 206 | 152
Not completed — Protocol Violation | 1 | 0
Not completed — No Study Treatment Given | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cabozantinib (XL184) | Placebo | Total
Number analyzed (Participants) | 470 | 237 | 707
Age, Continuous [Median (Full Range); unit: years] | 64.0 [22 to 86] | 64.0 [24 to 86] | 64.0 [22 to 86]
Age, Customized [Count of Participants; unit: Participants]
  Age, Customized: < 65 years old | 240 | 124 | 364
  Age, Customized: 65 to < 75 years old | 158 | 75 | 233
  Age, Customized: 75 to < 85 years old | 67 | 35 | 102
  Age, Customized: ≥ 85 years old | 5 | 3 | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 91 | 35 | 126
  Male | 379 | 202 | 581
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 18 | 12 | 30
  Not Hispanic or Latino | 417 | 215 | 632
  Unknown or Not Reported | 35 | 10 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 159 | 82 | 241
  Native Hawaiian or Other Pacific Islander | 3 | 0 | 3
  Black or African American | 8 | 11 | 19
  White | 264 | 130 | 394
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 36 | 13 | 49
Geographic Region [Count of Participants; unit: Participants]
  Australia / New Zealand | 15 | 11 | 26
  Asia | 116 | 59 | 175
  Europe | 231 | 108 | 339
  North America (USA / Canada) | 108 | 59 | 167
Presence of extrahepatic spread of disease and/or macrovascular invasion (stratification per IxRS) [Count of Participants; unit: Participants] — Interactive voice/web response system (IxRS)
  Participants
    Yes | 368 | 186 | 554
    No | 102 | 51 | 153
Etiology of disease (stratification factor per IxRS), [Count of Participants; unit: Participants]
  HBV (with or without known HCV) | 182 | 90 | 272
  HCV (without known HBV) | 100 | 51 | 151
  Other (neither HBV nor HCV) | 188 | 96 | 284
Geographic region (stratification factor per IxRS) [Count of Participants; unit: Participants]
  Asia | 116 | 59 | 175
  Other Regions | 354 | 178 | 532
Eastern Cooperative Oncology Group Performance Status (ECOG PS) [Count of Participants; unit: Participants] — The ECOG performance scale is:
  0 = Normal activity. Fully active, able to carry on all predisease performance without restriction, 1 = Symptoms, but ambulatory. Restricted in physically strenuous activity, but ambulatory and able to carry out work of a light or sedentary nature (eg, light housework, office work), 2 = In bed < 50% of the time. Ambulatory and capable of all self-care, but unable to carry out any work activities. Up and about more than 50% of waking hours.
  Participants
    0 | 245 | 131 | 376
    1 | 224 | 106 | 330
    2 | 1 | 0 | 1
Smoking history [Count of Participants; unit: Participants]
  Current | 78 | 42 | 120
  Former | 229 | 122 | 351
  Never | 160 | 71 | 231
  Missing | 3 | 2 | 5
Alcohol use [Count of Participants; unit: Participants]
  Current | 65 | 30 | 95
  Former | 223 | 124 | 347
  Never | 176 | 81 | 257
  Missing | 6 | 2 | 8
Weight [Median (Full Range); unit: kg] | 69 [35 to 130] | 71.5 [41 to 125] | 70.25 [35 to 130]
Body Mass Index (BMI) [Median (Full Range); unit: kg / m^2] | 24.1 [15 to 47] | 24.9 [17 to 42] | 24.5 [15 to 47]

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: The primary analysis of OS is defined as the time from randomization to death from any cause. The analysis was based on a second planned interim analysis prespecified to be performed at approximately the 75% information fraction (ie, at approximately 466 deaths). The data cutoff date for this event-driven analysis in the Intent to Treat (ITT) population was 01 June 2017. Median OS was calculated using the Kaplan-Meier estimates.
Time Frame: Up to 45 months
Population: The ITT population was used and included 707 randomized subjects (470 cabozantinib, 237 placebo) in the second interim analysis with a cutoff date of 01 June 2017.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib (XL184) | Placebo
Number analyzed (Participants) | 470 | 237
months | 10.2 [9.1 to 12.0] | 8.0 [6.8 to 9.4]
Statistical Analysis 1: Comparison: Cabozantinib (XL184) vs Placebo; Test type: Superiority; p = 0.0049, Log Rank; The Log-Rank Test was stratified by etiology of disease, geo. region, presence of extrahepatic spread of disease and/or macrovascular invasion; Hazard Ratio (HR) = 0.76, 95% CI 2-sided [0.63 to 0.92]

2. Secondary Outcome: Progression-Free Survival (PFS)
Description: Duration of PFS is defined as the time of randomization to the earlier of the following events, progressive disease as determined by Investigator (per RECIST 1.0, which is defined by a ≥ 20% increase in the sum of the longest diameter of target lesions from baseline) or death due to any cause. A Kaplan- Meier analysis was performed to estimate the median duration.
Time Frame: Up to 45 months
Population: The prespecified primary analysis of PFS was based on the first 707 randomized subjects (470 cabozantinib, 237 placebo).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cabozantinib (XL184) | Placebo
Number analyzed (Participants) | 470 | 237
months | 5.2 [4.0 to 5.5] | 1.9 [1.9 to 1.9]
Statistical Analysis 1: Comparison: Cabozantinib (XL184) vs Placebo; Test type: Superiority; p < 0.0001, Log Rank; The Log Rank Test was stratified by etiology of disease, geographic region, presence of extrahepatic spread of disease and/or macrovascular invasion; Hazard Ratio (HR) = 0.44, 95% CI 2-sided [0.36 to 0.52]

3. Secondary Outcome: Objective Response Rate (ORR)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: ORR is measured by radiologic assessment every 8 weeks after randomization until disease progression or discontinuation of study treatment (up to 45 months)
Population: The analysis of ORR was performed in the ITT population (all randomized: 470 cabozantinib, 237 placebo) based upon response determined by Investigator per RECIST 1.1
Measure: Count of Participants; unit: Participants
Arm/Group | Cabozantinib (XL184) | Placebo
Number analyzed (Participants) | 470 | 237
Participants | 18 | 1
Statistical Analysis 1: Comparison: Cabozantinib (XL184) vs Placebo; Test type: Superiority; p = 0.0086, Cochran-Mantel-Haenszel

ADVERSE EVENTS:
Time Frame: Up to 61 weeks
Description: The safety data includes subjects who were randomized and treated. Of 707 patients, 470 were randomized to received cabozantinib and 237 to placebo. Three subjects in the cabozantinib arm were randomized but did not receive study drug. Thus, a total of 704 subjects received study treatment in the Safety Population (467 cabozantinib, 237 placebo).
Arm/Group | Cabozantinib (XL184) | Placebo
All-Cause Mortality (participants affected / at risk) | 314/467 | 167/237
Serious Adverse Events (participants affected / at risk) | 232/467 | 87/237
Other Adverse Events (participants affected / at risk) | 445/467 | 173/237
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (XL184) (N=467) | Placebo (N=237)
Anaemia (Blood and lymphatic system disorders) | 4 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 0
Lymphopenia (Blood and lymphatic system disorders) | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 1 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 5 | 0
Acute myocardial infarction (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 1 | 0
Myocardial infarction (Cardiac disorders) | 0 | 1
Hypothyroidisim (Endocrine disorders) | 1 | 0
Retinal vein thrombosis (Eye disorders) | 1 | 0
Sudden visual loss (Eye disorders) | 1 | 0
Abdominal Pain (Gastrointestinal disorders) | 6 | 9
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Anal fistula (Gastrointestinal disorders) | 2 | 0
Ascites (Gastrointestinal disorders) | 12 | 3
Colitis (Gastrointestinal disorders) | 1 | 0
Constipation (Gastrointestinal disorders) | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 5 | 1
Duodenal perforation (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric perforation (Gastrointestinal disorders) | 2 | 0
Gastric varices haemorrhage (Gastrointestinal disorders) | 1 | 1
Gastritis erosive (Gastrointestinal disorders) | 1 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 4 | 1
Gastrointestinal ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Haematemesis (Gastrointestinal disorders) | 1 | 1
Ileus (Gastrointestinal disorders) | 1 | 0
Intestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Intestinal perforation (Gastrointestinal disorders) | 0 | 1
Large intestine perforation (Gastrointestinal disorders) | 2 | 0
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 2 | 0
Mesenteric atermy thrombosis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 1
Oesophageal varices haemorrhage (Gastrointestinal disorders) | 7 | 5
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Pancreatic pseudocyst (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 2 | 1
Pancreatitis acute (Gastrointestinal disorders) | 3 | 0
Peritoneal haemorrhage (Gastrointestinal disorders) | 0 | 1
Portal hypertensive gastropathy (Gastrointestinal disorders) | 1 | 0
Proctalgia (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 3 | 2
Rectal ulcer haemorrhage (Gastrointestinal disorders) | 0 | 1
Thrombosis mesenteric vessel (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 3 | 2
Vomiting (Gastrointestinal disorders) | 4 | 4
Asthenia (General disorders) | 9 | 0
Chest pain (General disorders) | 1 | 0
Death (General disorders) | 1 | 1
Fatigue (General disorders) | 6 | 1
General physical health deterioration (General disorders) | 17 | 8
Influenza like illness (General disorders) | 1 | 0
Infusion site extravasation (General disorders) | 1 | 0
Local swelling (General disorders) | 0 | 1
Multi-organ failure (General disorders) | 2 | 0
Non-cardiac chest pain (General disorders) | 1 | 0
Oedema (General disorders) | 2 | 0
Oedema peripheral (General disorders) | 3 | 0
Pain (General disorders) | 2 | 0
Pyrexia (General disorders) | 4 | 1
Acute hepatic failure (Hepatobiliary disorders) | 1 | 0
Bile duct obstruction (Hepatobiliary disorders) | 3 | 0
Bile duct stenosis (Hepatobiliary disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 3 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 1 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 1
Chronic hepatic failure (Hepatobiliary disorders) | 0 | 1
Dilatation intrahepatic duct acquired (Hepatobiliary disorders) | 0 | 1
Gallbladder perforation (Hepatobiliary disorders) | 1 | 0
Hepatic cirrhosis (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 8 | 8
Hepatic lesion (Hepatobiliary disorders) | 0 | 2
Hepatic pain (Hepatobiliary disorders) | 0 | 1
Hepatorenal syndrome (Hepatobiliary disorders) | 1 | 1
Hyperbilirubinaemia (Hepatobiliary disorders) | 2 | 1
Ischaemic hepatitis (Hepatobiliary disorders) | 1 | 0
Jaundice (Hepatobiliary disorders) | 0 | 2
Liver disorder (Hepatobiliary disorders) | 1 | 0
Portail vein thrombosis (Hepatobiliary disorders) | 3 | 0
Abscess jaw (Infections and infestations) | 1 | 0
Anal abscess (Infections and infestations) | 3 | 0
Bacteraemia (Infections and infestations) | 1 | 1
Biliary sepsis (Infections and infestations) | 0 | 2
Biliary tract infection (Infections and infestations) | 1 | 0
Bronchitis (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Cellulitis of male external genital organ (Infections and infestations) | 1 | 0
Clostridium dificile colitis (Infections and infestations) | 1 | 0
Clostridium dificile infection (Infections and infestations) | 1 | 1
Empyema (Infections and infestations) | 1 | 0
Gangrene (Infections and infestations) | 1 | 0
Gastroenteritis (Infections and infestations) | 2 | 1
Gastroenteritis viral (Infections and infestations) | 1 | 0
Gastroenteritis viral infection (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 1 | 0
Infection (Infections and infestations) | 1 | 1
Liver abscess (Infections and infestations) | 1 | 0
Lower respiratory tract infection (Infections and infestations) | 0 | 1
Lung infection (Infections and infestations) | 1 | 0
Peritonitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 16 | 6
Pneumonia bacterial (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 3 | 2
Sepsis syndrome (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 1 | 1
Staphylococcal sepsis (Infections and infestations) | 1 | 0
Subcutaneous abscess (Infections and infestations) | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 3 | 1
Urosepsis (Infections and infestations) | 1 | 0
Wound sepsis (Infections and infestations) | 1 | 0
Compression fracture (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0
Femur fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1
Intestinal anastomosis complication (Injury, poisoning and procedural complications) | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0
Multiple fractures (Injury, poisoning and procedural complications) | 1 | 0
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 | 1
Radius fracture (Injury, poisoning and procedural complications) | 1 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0
Amylase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 3 | 0
Blood bilirubin increased (Investigations) | 3 | 0
Blood creatine increased (Investigations) | 1 | 0
Gamma-glutamytransferase increased (Investigations) | 1 | 0
Lymphcyte count decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Oesophaggogastroduodenoscopy (Investigations) | 0 | 1
Oxygen saturation decreased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
Cachexia (Metabolism and nutrition disorders) | 1 | 0
Decreased appetite (Metabolism and nutrition disorders) | 4 | 0
Dehydration (Metabolism and nutrition disorders) | 4 | 2
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hyperammonaemia (Metabolism and nutrition disorders) | 0 | 1
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 2 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 5 | 0
Hypophagia (Metabolism and nutrition disorders) | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 2 | 1
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Intervertebral disc protusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Musculoskletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 | 0
Acute lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Head and neck cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 39 | 22
Intracranial tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Metastases to bone (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 3
Metastases to lung (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 | 0
Metastases to spine (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
Metastatic pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumor associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumor compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumor haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aphasia (Nervous system disorders) | 1 | 0
Cerebral haemorrhage (Nervous system disorders) | 1 | 0
Cerebral infarction (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 4 | 0
Cervicobrachial syndrome (Nervous system disorders) | 1 | 0
Convulsion (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Encephalopathy (Nervous system disorders) | 1 | 0
Hepatic encephalopathy (Nervous system disorders) | 15 | 1
Hyperammonaemic encephalopathy (Nervous system disorders) | 1 | 0
Ischaemic stroke (Nervous system disorders) | 2 | 0
Somnolence (Nervous system disorders) | 1 | 0
Spinal cord compression (Nervous system disorders) | 3 | 1
Syncope (Nervous system disorders) | 2 | 0
Completed suicide (Psychiatric disorders) | 1 | 0
Delirium (Psychiatric disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 1
Azotaemia (Renal and urinary disorders) | 0 | 1
Calculus ureteric (Renal and urinary disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Prerenal failure (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 1
Renal failure acture (Renal and urinary disorders) | 2 | 2
Pelvic pain (Reproductive system and breast disorders) | 1 | 1
Scrotal pain (Reproductive system and breast disorders) | 1 | 0
Testicular swelling (Reproductive system and breast disorders) | 1 | 0
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 2 | 3
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Oesophagobronchial fistula (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 | 2
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Diabetic ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia (Skin and subcutaneous tissue disorders) | 6 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Aneurysm (Vascular disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 2 | 0
Haematoma (Vascular disorders) | 1 | 0
Hypertension (Vascular disorders) | 2 | 1
Hypotension (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 1 | 0
Peripheral artery thrombosis (Vascular disorders) | 0 | 1
Peripheral ischaemia (Vascular disorders) | 1 | 0
Thrombosis (Vascular disorders) | 1 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
Respiratory crisis (verbatim) (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cabozantinib (XL184) (N=467) | Placebo (N=237)
Thrombocytopenia (Blood and lymphatic system disorders) | 51 | 1
Hypothyroidism (Endocrine disorders) | 38 | 1
Diarrhoea (Gastrointestinal disorders) | 251 | 43
Dyspepsia (Gastrointestinal disorders) | 47 | 7
Nausea (Gastrointestinal disorders) | 147 | 41
Stomatitis (Gastrointestinal disorders) | 63 | 5
Vomiting (Gastrointestinal disorders) | 118 | 24
Asthenia (General disorders) | 99 | 17
Fatigue (General disorders) | 209 | 70
Mucosal inflammation (General disorders) | 65 | 5
Alanine aminotransferase increased (Investigations) | 79 | 13
Aspartate aminotransferase increased (Investigations) | 103 | 27
Platelet count decreased (Investigations) | 45 | 7
Weight decreased (Investigations) | 80 | 14
Decreased appetite (Metabolism and nutrition disorders) | 224 | 43
Hypoalbuminaemia (Metabolism and nutrition disorders) | 55 | 12
Hypokalaemia (Metabolism and nutrition disorders) | 44 | 4
Hypomagnesaemia (Metabolism and nutrition disorders) | 29 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 39 | 4
Pain in extremity (Musculoskeletal and connective tissue disorders) | 44 | 9
Dysgeusia (Nervous system disorders) | 56 | 5
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 90 | 5
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 217 | 12
Rash (Skin and subcutaneous tissue disorders) | 58 | 14
Hypertension (Vascular disorders) | 137 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreements with investigators vary; constant is our right to review results communications prior to public release, and embargo communications for a period of ≤ 60 days from submittal for review. We do not prohibit investigators from publishing, but we may require previously undisclosed confidential information, other than study results, to be removed from publications, and single-center publications are postponed until after publication of the trial's primary multicenter publication.

DOCUMENTS (2):
  • Study Protocol (2016-07-12): https://cdn.clinicaltrials.gov/large-docs/26/NCT01908426/Prot_000.pdf
  • Statistical Analysis Plan (2016-06-08): https://cdn.clinicaltrials.gov/large-docs/26/NCT01908426/SAP_001.pdf